CLINICAL TRIAL: NCT01725152
Title: A Controlled, Double-blind, Crossover Trial of Ganaxolone in Children With Fragile X Syndrome
Brief Title: Ganaxolone Treatment in Children With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Collaborators: University of California, Davis (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-0800
Record Dates: First submitted 2012-11-07; First posted 2012-11-12 (Estimated); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Fragile x Syndrome
Keywords: fragile x syndrome; ganaxolone; anxiety; attention; pediatric
MeSH Terms: conditions — Fragile X Syndrome; Anxiety Disorders | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ganaxolone then Placebo (Experimental): Participants first received ganaxolone. They were first titrated up to the 12 milligram per kilogram (mg/kg) three times daily (tid) during a 2-week titration phase, then maintained on that dose for an additional 4 weeks. After a washout period of 2 weeks, participants received placebo for a duration of 6 weeks (from week 8 to 14).
  Interventions: Drug: Ganaxolone; Drug: Placebo
- Placebo then Ganaxolone (Experimental): Participants first received placebo. They were first titrated up to the 12 mg/kg tid during a 2-week titration phase, then maintained on that dose for an additional 4 weeks. After a washout period of 2 weeks, participants received ganaxolone for a duration of 6 weeks (from week 8 to 14).
  Interventions: Drug: Ganaxolone; Drug: Placebo

INTERVENTIONS:
Drug: Ganaxolone — oral suspension, given in 3 divided doses
Drug: Placebo — oral suspension, given in 3 divided doses

SUMMARY:
This Phase 2 proof-of-concept study is a double-blind, randomized, placebo-controlled, crossover study to investigate ganaxolone treatment in children with fragile x syndrome (FXS). The objective of the study is to assess the safety, tolerability and efficacy of ganaxolone in the treatment of anxiety and attention in subjects with FXS.

DETAILED DESCRIPTION:
This is a single center study conducted at University of California Davis (UCD) MIND Institute. Children with FXS between the ages of 6-17 years, inclusive will be randomized at a 1:1 ratio to receive ganaxolone or placebo treatment for 6 weeks, discontinue treatment and washout for 2 weeks, and then cross over to the opposite treatment for another 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* molecular documentation of FMR1 full mutation
* ages 6-17 yrs, inclusive
* sexually active subjects are required to use a medically acceptable form of birth control

Exclusion Criteria:

* non-English or Spanish speaking subjects
* concomitant systemic steroid, vigabatrin, felbamate and ketoconazole
* changes in medications within last 2 months
* clinically unstable medical disease, progressive CNS disease/disorder
* history of recurrent status epilepticus
* unwilling to withhold grapefruit or grapefruit juice for the duration of the study
* actively suicidal

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10-16 (Actual); Study Completion 2016-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- M.I.N.D. Institute at University of California at Davis Medical Center, Sacramento, California, United States
- Antwerp University Hospital, Edegem, Belgium

REFERENCES:
- [Derived] Ligsay A, Van Dijck A, Nguyen DV, Lozano R, Chen Y, Bickel ES, Hessl D, Schneider A, Angkustsiri K, Tassone F, Ceulemans B, Kooy RF, Hagerman RJ. A randomized double-blind, placebo-controlled trial of ganaxolone in children and adolescents with fragile X syndrome. J Neurodev Disord. 2017 Aug 2;9(1):26. doi: 10.1186/s11689-017-9207-8. PMID 28764646

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 participants from the University of California at Davis Medical Center site and 11 participants from a Belgium site between November 1, 2012 and November 1, 2016 were enrolled in the study.
Pre-assignment Details: 59 participants were randomized in the study.
Groups:
- Ganaxolone, Then Placebo: Participants received ganaxolone were first titrated up to the 12 milligram per kilogram (mg/kg) three times daily (tid) during a 2-week titration phase, then maintained on that dose for an additional 4 weeks. After a washout period of 2 weeks, they received placebo for a duration of 6 weeks (from week 8 to 14).
- Placebo, Then Ganaxolone: Participants received placebo were first titrated up to the 12 mg/kg tid during a 2-week titration phase, then maintained on that dose for an additional 4 weeks. After a washout period of 2 weeks, they received ganaxolone for a duration of 6 weeks (from week 8 to 14).
Period: Treatment Period 1 (Week 1 to Week 6)
Arm/Group | Ganaxolone, Then Placebo | Placebo, Then Ganaxolone
Started | 30 | 29
Completed | 26 | 29
Not Completed | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Consent Withdrawn | 1 | 0
Period: Washout Period (2 Weeks)
Arm/Group | Ganaxolone, Then Placebo | Placebo, Then Ganaxolone
Started | 26 | 29
Completed | 26 | 29
Not Completed | 0 | 0
Period: Treatment Period 2 (Week 8 to Week 14)
Arm/Group | Ganaxolone, Then Placebo | Placebo, Then Ganaxolone
Started | 26 | 29
Completed | 25 | 26
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who have taken at least one dose of study drug in Treatment period 1.
Groups:
- Ganaxolone, Then Placebo: Participants received ganaxolone were first titrated up to the 12 mg/kg tid during a 2-week titration phase, then maintained on that dose for an additional 4 weeks. After a washout period of 2 weeks, they received placebo for a duration of 6 weeks (from week 8 to 14).
- Total: Total of all reporting groups
Arm/Group | Ganaxolone, Then Placebo | Placebo, Then Ganaxolone | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.58 (3.245) | 11.33 (3.368) | 10.95 (3.299)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 27 | 23 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 22 | 23 | 45
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Improvement (CGI-I) Scale
Description: The CGI-I scale is a clinician-rated 7-point scale used to assess how much the participant's illness had improved or worsened relative to a Baseline state at the beginning of the intervention. It was rated as: 1. "very much improved"; 2. "much improved"; 3. "minimally improved"; 4. "no change"; 5. "minimally worse"; 6. "much worse"; 7. "very much worse". Higher scores indicated worse condition.
Time Frame: Week 14 (End of Treatment)
Population: Intention-to-Treat (ITT) Population consisted of all participants who received medication and who had at least one post-Baseline assessment. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Ganaxolone: Participants who received Ganaxolone up to 12 mg/kg tid in the first 6 weeks or last 6 weeks of the study.
- Placebo: Participants who received placebo (matching Ganaxolone) in the first 6 weeks or last 6 weeks of the study.
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 52 | 54
Scores on a scale | 3.4 (0.13) | 3.5 (0.13)
Statistical Analysis 1: Comparison: Ganaxolone vs Placebo; Null hypothesis of no treatment difference in CGI-I will be assessed using a linear mixed-effects model for repeated measures, accounting for treatment (ganaxolone versus placebo) and period at a significant level of 0.05. A sample size of 30 participants in each arm/group was planned in the study will have 90% power to detect a modest effect size of 0.6 at level 0.05 in CGI-I. With a possible dropout rate of 15%, the power for testing the effect size becomes 84%; Test type: Superiority; p = 0.4475, Linear mixed-effect

2. Secondary Outcome: Pediatric Anxiety Rating Scale (PARS) Total Score
Description: Pediatric Anxiety Rating Scale (PARS) is a clinician administered measure of anxiety in children and adolescents. The PARS is comprised of a 50-item symptom checklist used to determine the presence or absence of specific anxiety symptoms during the prior week and 7 severity/impairment items, each scored from 0 to 5. The score on the 7 items allows the clinician to rate symptom severity and associated impairment on a range from 0 to 35, with higher scores reflecting greater symptom severity and associated impairment.
Time Frame: Week 14 (End of Treatment)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 52 | 54
Scores on a scale | 8.3 (0.54) | 9.2 (0.54)

3. Secondary Outcome: Visual Analogue Scale (VAS)
Description: A semi-structured VAS design was employed, providing two of the three behaviors to be assessed as anxiety and attention, chosen by caregiver(s) of one additional behavior from a bank of five. This bank included sociability, attention, aggression, language, and hyperactivity/impulsivity. Parents mark on a visual line measuring 10 centimeters (cm) with "worst behavior" at 0 cm and "best behavior" at 10 cm. For each behavior the caregiver is instructed to mark their impression of behavior at Baseline visit and again at each visit. The calculated distance in cm between the baseline and each visit marks thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the least square mean distance and its corresponding standard error in cm from the "worst behavior" side, at baseline. Smaller the value, worser the behavior.
Time Frame: Week 14 (End of Treatment)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Centimeters (cm)
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 51 | 54
Centimeters (cm)
  Severity of Anxiety | 5.6 (0.27) | 5.0 (0.26)
  Severity of Attention | 4.4 (0.24) | 3.9 (0.24)
  Severity of Target Behavior 3 | 4.4 (0.28) | 3.9 (0.27)

4. Secondary Outcome: Anxiety, Depression, and Mood Scale (ADAMS)
Description: The ADAMS is a 28-item behavior-based informant instrument rated by the parent(s), legal authorized guardian(s), or consistent caregiver(s). The scale is composed of 5 factors, which addresses Manic/Hyperactive Behavior, Depressed Mood, Social Avoidance, General Anxiety, and Obsessive/Compulsive Behavior. Items are scored on a 0-3 Likert scale that combines frequency and severity ratings (where 0=behavior has not occurred or is not a problem, 3=behavior occurs a lot or is a severe problem). Each subscale score is calculated separately; the scale range for Manic/Hyperactive Behavior is 0-15; for Depressed Mood, 0-21; for Social Avoidance, 0-21; for General Anxiety, 0-21; for Obsessive Behavior, 0-9. There is an overlapped item between Manic/Hypertension Behavior and General Anxiety; hence, the subscale ranges appear to reflect scores for 29 items instead of 28 items.
Time Frame: Week 14 (End of Treatment)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 50 | 54
Scores on a scale
  Manic/Hyperactive Behavior Total | 7.4 (0.42) | 7.8 (0.40)
  Depress Mood Total: number analyzed (Participants) | 49 | 54
  Depress Mood Total | 3.5 (0.32) | 2.6 (0.32)
  Social Avoidance Total | 5.8 (0.42) | 6.3 (0.41)
  General Anxiety Total: number analyzed (Participants) | 50 | 53
  General Anxiety Total | 6.2 (0.45) | 7.0 (0.44)
  Obsessive/Compulsive Behavior Total | 2.7 (0.21) | 2.8 (0.20)

5. Secondary Outcome: Aberrant Behavior Checklist (ABC)
Description: The ABC is a 58-item parent rated from 0 (not at all a problem) to 3 (the problem is severe in degree with 6 subscales: Irritability (includes agitation, aggression, and self-injury, 15 items) with range of scores from 0-45; Social Withdrawal/Lethargy (16 items) with range of scores from 0-48; Stereotypy (7 items) with range of scores from 0-21; Hyperactivity (16 items) with range of scores from 0-48; Inappropriate Speech (4 items) with range of scores from 0-12 and Social avoidance (4 items) with range of scores from 0-12. Higher scores indicated greater severity. Social Withdrawal and Lethargy are reporting the same scale and Social Avoidance is a subscale of Social Withdrawal; hence, the subscale ranges appear to reflect scores for 62 items instead of 58 items.
Time Frame: Week 14 (End of Treatment)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 50 | 54
Scores on a scale
  Total - Subscale I (Irritability): number analyzed (Participants) | 49 | 53
  Total - Subscale I (Irritability) | 15.7 (0.87) | 16.1 (0.86)
  Total - Subscale II (Social Withdrawal/Lethargy): number analyzed (Participants) | 50 | 53
  Total - Subscale II (Social Withdrawal/Lethargy) | 5.6 (0.53) | 5.7 (0.54)
  Total - Subscale III - (Stereotypy) | 5.7 (0.40) | 6.4 (0.39)
  Total - Subscale IV (Hyperactivity) | 11.3 (0.65) | 12.3 (0.62)
  Total - Subscale V (Inappropriate Speech) | 5.1 (0.32) | 5.3 (0.31)
  Total - Subscale VI (Social Avoidance) | 2.4 (0.22) | 2.8 (0.21)

6. Secondary Outcome: Swanson, Nolan, and Pelham-IV Questionnaire (SNAP-IV)
Description: The SNAP-IV is a revision of the Swanson, Nolan, and Pelham (SNAP) Questionnaire. The SNAP-IV: ADHD Inattention Subscale (items 1-9) scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). Possible scores ranged from 0-27; higher scores indicated a greater intensity. The SNAP-IV ADHD Hyperactivity/Impulsivity Subscale (items 10-18) scores the intensity of each item in the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). Possible scores ranged from 0-27; higher scores indicated a greater intensity. SNAP-IV ADHD Combined Scale score (inattention + hyperactivity/impulsivity) ranged from 0-54. A low score of 0 indicates less inattention + hyperactivity/impulsivity. A high score of 54 indicates more inattention + hyperactivity.
Time Frame: Week 14 (End of Treatment)
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 50 | 53
Scores on a scale
  ADHD Inattention | 15.5 (0.66) | 14.6 (0.62)
  ADHD Hyperactivity/Impulsive | 13.9 (0.66) | 12.6 (0.64)
  ADHD Combined | 29.3 (1.19) | 27.1 (1.14)

ADVERSE EVENTS:
Time Frame: Up to 14 Weeks
Description: Safety Population included all participants who received at least one dose of intervention. One participant mistakenly did not cross over to receive placebo and remained on Ganaxolone during Period 2 as a result of a pharmacy error.
Arm/Group | Ganaxolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/54
Other Adverse Events (participants affected / at risk) | 49/59 | 46/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=59) | Placebo (N=54)
Fatigue (General disorders) | 29 | 11
Condition aggravated (General disorders) | 10 | 6
Somnolence (Nervous system disorders) | 20 | 3
Headache (Nervous system disorders) | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 7
Vomiting (Gastrointestinal disorders) | 8 | 5
Upper respiratory tract infection (Infections and infestations) | 9 | 11
Agitation (Psychiatric disorders) | 3 | 8
Aggression (Psychiatric disorders) | 6 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 8 | 2
Pyrexia (General disorders) | 1 | 3
Irritability (General disorders) | 1 | 2
Thirst (General disorders) | 1 | 1
Hyperpyrexia (General disorders) | 0 | 1
Hypersomnia (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 2 | 1
Coordination abnormal (Nervous system disorders) | 1 | 1
Poor quality sleep (Nervous system disorders) | 2 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 1
Repetitive speech (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Drooling (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 1 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4
Rhinitis (Infections and infestations) | 2 | 2
Otitis media (Infections and infestations) | 1 | 1
Candida nappy rash (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0
Emotional disorder (Psychiatric disorders) | 1 | 2
Self injurious behaviour (Psychiatric disorders) | 1 | 2
Stereotypy (Psychiatric disorders) | 3 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 1 | 1
Terminal insomnia (Psychiatric disorders) | 0 | 2
Tic (Psychiatric disorders) | 2 | 0
Affect lability (Psychiatric disorders) | 0 | 1
Binge eating (Psychiatric disorders) | 0 | 1
Dysphemia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Negativism (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Obsessive thoughts (Psychiatric disorders) | 0 | 1
Sleep talking (Psychiatric disorders) | 1 | 1
Staring (Psychiatric disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 1
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tooth avulsion (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Incontinence (Renal and urinary disorders) | 0 | 1
Ketonuria (Renal and urinary disorders) | 0 | 1
Aortic dilatation (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Pallor (Vascular disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Nipple swelling (Reproductive system and breast disorders) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 1
Blepharitis (Eye disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Treatment noncompliance (Social circumstances) | 0 | 1
Dental operation (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No